CLINICAL TRIAL: NCT07353073
Title: A Prospective, Single-Arm, Phase II Clinical Study of Neoadjuvant Therapy With Pucotenlimab, Lenvatinib, and Temozolomide for Resectable Head and Neck Mucosal Melanoma (PLT-NAT-HNMM-II)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH9H-2025-T534-1
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Mucosal Melanomas
Keywords: head and neck mucosal melanoma; pucotenlimab
MeSH Terms: interventions — lenvatinib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pucotenlimab in combination with lenvatinib and temozolomide (Experimental): Preoperatively, patients will receive 2 cycles of pucotenlimab (200 mg every 3 weeks, or 3 mg/kg every 3 weeks) combined with lenvatinib (20 mg once daily) and temozolomide (150 mg/m² orally once daily for 5 consecutive days per 28-day cycle). Postoperatively, treatment with pucotenlimab will be continued until a total of 1 year of therapy is completed.
  Interventions: Drug: Preoperatively, patients will receive 2 cycles of pucotenlimab (200 mg every 3 weeks, or 3 mg/kg every 3 weeks) combined with lenvatinib (20 mg once daily) and temozolomide (150 mg/m² orally once dail

INTERVENTIONS:
Drug: Preoperatively, patients will receive 2 cycles of pucotenlimab (200 mg every 3 weeks, or 3 mg/kg every 3 weeks) combined with lenvatinib (20 mg once daily) and temozolomide (150 mg/m² orally once dail — Preoperatively, patients will receive 2 cycles of pucotenlimab (200 mg every 3 weeks, or 3 mg/kg every 3 weeks) combined with lenvatinib (20 mg once daily) and temozolomide (150 mg/m² orally once daily for 5 consecutive days per 28-day cycle). Postoperatively, treatment with pucotenlimab will be continued until a total of 1 year of therapy is completed.

SUMMARY:
This study aims to conduct a prospective clinical trial investigating the use of pucotenlimab in combination with lenvatinib and temozolomide as neoadjuvant and postoperative adjuvant therapy for resectable oral and head and neck mucosal melanoma. The primary objectives are to evaluate the safety and efficacy of this combination regimen in the neoadjuvant treatment of head and neck mucosal melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years, regardless of gender.
* Histologically confirmed primary, resectable Head and Neck Mucosal Melanoma (HNMM), with measurable lesions (spiral CT scan ≥10 mm, meeting RECIST 1.1 criteria) or intraoral patch lesions deemed evaluable by the study investigators.
* ECOG performance status of 0 or 1.
* Life expectancy ≥12 weeks.
* At least one measurable lesion according to RECIST 1.1 criteria. Previously treated lesions can also serve as target lesions if disease progression has occurred.
* Availability of tumor tissue for PD-L1 testing (paraffin-embedded specimens from within the last 2 years or fresh tumor tissue).
* Organ function must meet the following requirements (within 14 days prior to the first dose of the study drug):
* **Bone Marrow:** Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L, platelet count (PLT) ≥100 × 10⁹/L, hemoglobin (HB) ≥9 g/dL (no blood transfusion or blood product administration within 14 days prior to testing).
* **Liver:** Serum total bilirubin (TBIL) ≤1.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN (if liver metastases are present, AST and ALT ≤5 × ULN are permitted).
* **Kidneys:** Serum creatinine ≤1.5 × ULN or creatinine clearance ≥60 mL/min, blood urea nitrogen ≤200 mg/L.
* Thyroid-stimulating hormone (TSH) ≤1 × ULN (if abnormal, free T3 [FT3] and free T4 [FT4] levels should also be assessed; if FT3 and FT4 levels are normal, the patient may be enrolled).
* Urine protein ≤1+; if urine protein >1+, a 24-hour urine protein collection is required, and the total amount must be ≤1 gram.
* Normal cardiac function, defined as an electrocardiogram (ECG) without clinically significant abnormalities and a left ventricular ejection fraction (LVEF) >50% as shown by echocardiography.
* Female subjects of childbearing potential must have a negative serum pregnancy test result prior to the first dose of the investigational drug.
* Male or female subjects of childbearing potential must use highly effective contraception methods (e.g., oral contraceptives, intrauterine devices, sexual abstinence, or barrier methods combined with spermicide) throughout the entire trial period and continue contraception for 90 days after the end of treatment.
* Subjects must voluntarily join the study, sign an informed consent form, demonstrate good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Prior treatment with PD-1/PD-L1/PD-L2/CTLA-4 antibodies, or drugs targeting T-cell receptor activation or inhibition (e.g., OX40, CD137).
2. Allergy to recombinant humanized anti-PD-1 monoclonal antibody or its components.
3. Cutaneous melanoma, ocular melanoma, or melanoma of unknown primary origin.
4. Primary lesion cannot be completely resected; presence of distant metastases; or local lesions are not indicated for surgery.
5. Concurrently receiving any other anti-tumor therapy.
6. Pregnancy, lactation, or women of childbearing potential not using contraception.
7. Uncontrolled severe acute infection.
8. Presence of any uncontrolled clinical condition, including but not limited to:

   * Persistent or active (severe) infection;
   * Poorly controlled diabetes;
   * Cardiac disease (NYHA Class III/IV congestive heart failure or heart block);
   * Current or suspected autoimmune disease, or history of autoimmune disease or syndromes requiring systemic steroid/immunosuppressant therapy, such as hypophysitis, colitis, hepatitis, nephritis, hyperthyroidism, hypothyroidism, etc.;
   * Occurrence of any of the following within 6 months prior to the first dose: deep vein thrombosis or pulmonary embolism; myocardial infarction; severe or unstable arrhythmia or angina; percutaneous coronary intervention, acute coronary syndrome, or coronary artery bypass graft; cerebrovascular accident, transient ischemic attack, or cerebral embolism.
9. Patients with active hepatitis B or C:

   * If HBsAg or HBcAb is positive, HBV DNA must be tested (excluded if above the upper limit of normal).
   * If HCV antibody is positive, HCV RNA must be tested (excluded if above the upper limit of normal).
10. Occurrence of any of the following within 6 months prior to the first dose: deep vein thrombosis or pulmonary embolism; myocardial infarction; severe or unstable arrhythmia or angina; percutaneous coronary intervention, acute coronary syndrome, or coronary artery bypass graft; cerebrovascular accident, transient ischemic attack, or cerebral embolism.
11. Any other severe, acute, or chronic medical condition or laboratory abnormality that, in the investigator's judgment, may increase study-related risk or potentially interfere with the interpretation of study results.
12. History of stem cell or organ transplantation.
13. History of psychoactive drug abuse with inability to abstain, or history of psychiatric disorders.
14. Patients whom the investigator judges to have poor compliance or other conditions making them unsuitable for participation in this trial.
15. Concurrent participation in other clinical studies, except for observational studies or those deemed non-conflicting with this study.
16. History of other malignancies within the past 5 years, except for cured basal cell carcinoma, squamous cell carcinoma of the skin, early-stage prostate cancer, and carcinoma in situ of the cervix.
17. Patients using immunosuppressants or systemic corticosteroids for immunosuppressive purposes (equivalent to >10mg/day prednisone) and continuing such use within 2 weeks prior to enrollment.
18. Patients who have received hematopoietic growth factors (e.g., G-CSF, erythropoietin) within 1 week prior to the first dose of the study drug.
19. Any underlying medical condition that, in the investigator's opinion, would increase the risk of study drug administration or confound the assessment of toxicity or adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Response Rate (pCR + Near-pCR + pPR). | Preoperatively, within 2-4 weeks after completing neoadjuvant therapy
  pCR (Pathological Complete Response, no residual tumor), near-pCR (Near Pathological Complete Response, tumor residue ≤10%), pPR (Pathological Partial Response, 10% < tumor residue ≤50%), and pNR (Pathological No Response, tumor residue >50%).

SECONDARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | Preoperatively, within 2-4 weeks after completing neoadjuvant therapy
  Defined as the proportion of subjects with no viable tumor cells in the postoperative resection specimen.
objective response rate | 4-8 weeks
  It refers to the proportion of patients whose tumor volume reduction, according to recognized response evaluation criteria (such as RECIST version 1.1 for solid tumors), meets predefined criteria and is maintained for a minimum required duration. This is the sum of the rates of complete response (CR) and partial response (PR).
adverse event (AE) | 1 year
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical trial participant administered a medicinal product, which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the product.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No